CLINICAL TRIAL: NCT00612638
Title: Phase I Trail of Temodar Plus O6-Benzylguanine (O6-BG) (NSC 637037) Plus Irinotecan (CPT-11) (NSC 616348) in the Treatment of Patients With Recurrent / Progressive Cerebral Anaplastic Gliomas
Brief Title: Ph. I Temozolomide + O6-BG + Irinotecan in Treatment of Pts w Recurrent / Progressive Cerebral Anaplastic Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Keryx / AOI Pharmaceuticals, Inc. (Industry); Pharmacia (Industry)
Responsible Party: David A. Reardon, MD, Duke University Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007681
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2009-01

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Temodar; Temozolomide; O6-Benzylguanine; O6-BG; NSC 637037; Irinotecan; CPT-11; Recurrent cerebral anaplastic glioma; Progressive cerebral anaplastic glioma; Malignant glioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — Temozolomide; O(6)-benzylguanine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pts receiving Dilantin, Tegretol or Phenobarbital
  Interventions: Drug: Temodar, O6-BG, and Irinotecan
- 2 (Experimental): Pts on anti-convulsants other than Dilantin, Tegretol / Phenobarbital / pts not on any anti-convulsants
  Interventions: Drug: Temodar, O6-BG, and Irinotecan

INTERVENTIONS:
Drug: Temodar, O6-BG, and Irinotecan — 2 separate strata accrued independently: Stratum 1-pts receiving Dilantin, Tegretol or phenobarbital. Stratum 2-pts on anti-convulsants other than Dilantin, Tegretol/phenobarbital/pts not on any anti-convulsants. O6-BG administered intravenously 120mg/m2, over 1hr, prior to administration of Temozolomide on day 1 of 21day cycle. O6-BG administered intravenously 30mg/m2/day, over 48hrs, immediately after completion of CPT-11 infusion on day 1 of 21-day cycle. Temozolomide administered orally 355mg/m2 within 60 mins of end of 1hr O6-BG infusion. Treatment cycles may be repeated every 3wks following dose of Temozolomide from previous cycle. CPT-11 administered intravenously in fasting state over 90mins. CPT-11 infusion will begin 1hr after Temozolomide administration. Initial doses 60mg/m2 for stratum 1 & 40mg/m2 for stratum2. Treatment cycles repeated every 3 wks following dose of CPT-11 from previous cycle.
  Other Names: Temodar-Temozolomide; O6-Benzylguanine-O6-BG; Irinotecan-Camptosar-CPT 11

SUMMARY:
Objectives:

To determine maximum tolerated dose of CPT-11 when administered following Temodar plus O6-benzylguanine To characterize any toxicity associated w combo of CPT-11 + Temodar plus O6-BG To observe pts for clinical antitumor response when treated w combo of CPT-11 + Temodar + O6-BG

DETAILED DESCRIPTION:
Objectives of study: to determine maximum tolerated dose of CPT-11 when administered following Temodar + O6-benzylguanine (O6-BG); to characterize any toxicity associated w combo of CPT-11 + Temodar + O6-BG; to observe pts for clinical antitumor response when treated w combo of CPT-11 + Temodar plus O6-BG. Pts have histologically confirmed diagnosis of recurrent primary malignant glioma. 2 separate strata accrued independently of each other: Stratum 1-pts receiving Dilantin, Tegretol/phenobarbital. Stratum 2-pts on anti-convulsants other than Dilantin, Tegretol/phenobarbital/pts not on any anti-convulsants. Each strata will be treated & escalated independent of each other.

Pre-chemo, O6-BG administered intravenously at 120 mg/m2, over 1hr, prior to administration of Temodar on day 1 of 21-day cycle. Post-chemo, O6-BG administered intravenously at 30 mg/m2/day, over 48hrs, immediately after completion of the CPT-11 infusion on day 1 of 21-day cycle. Temodar administered orally at 355 mg/m2, in fasting state, within 60 minutes of the end of 1hr O6-BG infusion. Treatment cycles may be repeated every 3 weeks following dose of Temozolomide from previous cycle. CPT-11 will be administered intravenously in fasting state over 90min. CPT-11 infusion will begin 1hr after Temozolomide administration. Initial doses 60 mg/m2 for stratum 1 & 40 mg/m2 for stratum 2. Treatment cycles may be repeated every 3 wks following dose of CPT-11 from previous cycle.

Major toxicities associated w CPT- 11 are myelosuppression & diarrhea. Temozolomide has been well tolerated by both adults & children w most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea & vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, & hepatotoxicity. Hypersensitivity reactions have not yet been noted w Temozolomide. As is case w many anti-cancer drugs, Temozolomide may be carcinogenic. O6-BG toxicities include transient lymphopenia has been seen w O6-BG as single agent. O6-BG in combo w other agents could cause exacerbation of any adverse event currently known to be caused by other agent,/ combo may result in events never previously associated w either agent. Animal studies indicated that agitation, lethargy, convulsions, nausea, vomiting, rapid heart rate, elevated liver functions, leukopenia, lymphopenia could be seen.

ELIGIBILITY:
Inclusion Criteria:

* Pts have histologically confirmed diagnosis of recurrent primary malignant glioma
* Age >18yrs
* Evidence of measurable recurrent/residual primary CNS neoplasm on contrast-enhanced MRI, unless medically contraindicated
* An interval of >2 wks between prior surgical resection/6 wks between prior XRT/chemo, & enrollment on protocol, unless there is unequivocal evidence of tumor progression after surgery, XRT/chemo
* KPS>60 percent
* Adequate hematologic, renal & liver function as demonstrated by lab values performed within 14 days, inclusive, prior to administration of chemo:
* ANC >1500/mm3
* Platelet count > 00,000/mm3
* Hemoglobin > 10gm/dL
* BUN & serum creatinine <1.5 x ULN
* Total serum bilirubin <1.5 x ULN
* SGOT & SGPT < 2.5 x ULN
* Alkaline phosphatase of< 2 x ULN
* Pts must have recovered from any effects of major surgery.=
* Pts must have life expectancy of >12wks
* Pts/legal guardian must give written, informed consent

Exclusion Criteria:

* Pts requiring immediate XRT
* Pts have not recovered from surgery
* Pts are not neurologically stable for 2wks prior to study entry
* Pts are poor medical risks because of non-malignant systemic disease as well as those w acute infection treated w intravenous antibiotics
* Frequent vomiting/medical condition that could interfere w oral medication intake
* Previous active malignancy treated in past year except for localized in-situ carcinomas & basal/squamous cell carcinoma of skin
* Known HIV positivity/AIDS-related illness
* Pregnant/nursing women
* Women of childbearing potential who are not using effective method of contraception. Women of childbearing potential must have negative serum pregnancy test 24 hrs prior to administration of study drug & be practicing medically approved contraceptive precautions
* Men who are not advised to use effective method of contraception
* Prior failure of CPT-11
* Pts taking immuno-suppressive agents other than prescribed corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities | 6 months

SECONDARY OUTCOMES:
Response rate & progression-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/